CLINICAL TRIAL: NCT02459210
Title: CLUES (Cognition for Learning and for Understanding Everyday Social Situations): An Adaptation of Cognitive Enhancement Therapy for Persons at Clinical High Risk for Psychosis
Brief Title: Adaptation of Cognitive Enhancement Therapy for Persons at Clinical High Risk for Psychosis
Acronym: CLUES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Matcheri S. Keshavan MD, Stanley Cobb Professor of Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014P000285; 1R34MH105596-01 (NIH)
Record Dates: First submitted 2015-04-14; First posted 2015-06-02 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Psychosis
Keywords: clinical high risk for psychosis; psychosis prodrome; cognitive remediation; psychosis prevention
MeSH Terms: conditions — Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLUES (Experimental): active treatment
  Interventions: Behavioral: CLUES
- therapy and computer games (Active Comparator): supportive therapy + computer games
  Interventions: Behavioral: therapy and computer games

INTERVENTIONS:
Behavioral: CLUES — Cognition for learning and for understanding everyday social situations intervention described above
  Arms: CLUES
Behavioral: therapy and computer games — Weekly psychotherapy+ computer games such as sporcle
  Arms: therapy and computer games

SUMMARY:
The purpose of this study is to test the feasibility of a modification of CET (Cognitive Enhancement Therapy) to address symptomatic and functional difficulties associated with Clinical High Risk for Psychosis (CHR).

Cognition for Learning and for Understanding Everyday Social Situations (CLUES) is designed to improve cognitive functioning (e.g., memory, attention, planning, etc.) in order to improve school, work, and social functioning. CLUES includes the following:

1. Computerized cognitive remediation ("exercises") to improve cognition.
2. Social-cognitive skills group designed to teach participants to act wisely in social situations.
3. Individual coaching sessions designed to enhance translation of skills learned from computer exercises and the group into real life.

CLUES is based on Hogarty and Greenwald's Cognitive Enhancement Therapy (CET), which was designed for treating individuals with schizophrenia. Research on CET for individuals with schizophrenia has found that CET appears to have helped participants improve cognition and social and work functioning.

This study will investigate the feasibility of CLUES for young people who are showing signs of clinical risk for psychosis.

Part 1: Preliminary open label trial of CLUES (n=8) to examine preliminary evidence of target engagement (change in cognition and social cognition), to refine assessment and recruitment approaches, to further optimize the treatment manual, and to ascertain feasibility and tolerability.

Part 2: Preliminary randomized controlled trial of CLUES vs supportive therapy (ST) + computer games to explore preliminary evidence of efficacy of CLUES vs. the control treatment (n=30).

DETAILED DESCRIPTION:
Psychotic disorders such as schizophrenia (SZ) are among the most disabling conditions in all of medicine. These disorders typically begin in adolescence or young adulthood, and are preceded by premorbid impairments in cognitive and social function dating from early childhood; these deficits worsen in adolescence and are accompanied by sub-threshold positive and negative symptoms (the prodromal, or clinical high risk state, CHR) before onset of the first psychotic episode. Recent staging models have operationalized approaches to defining early and late phases of CHR; Early CHR (stage 1a) is characterized by cognitive impairments and sub-threshold negative symptoms, while late CHR (stage 1b) is associated with sub-threshold positive and disorganized symptoms as well as further cognitive and functional declines. The emergence of cognitive and functional decline in Individuals at CHR who convert to psychosis highlights the importance of early intervention.

Impairments in cognition are present in children who later go on to develop SZ. Impairments in cognition are key rate-limiting factors to functional recovery from psychotic disorders and include deficits in psychomotor speed, memory, attention, reasoning, and social cognition. The latter include deficits in perspective-taking, emotion perception and regulation, clearly linked to functional outcome in SZ. Perspective-taking (ability to understand the thoughts, feelings, and intentions of others) and emotion regulation (ability to have cognitive control over emotional stimuli) are critical for healthy social development; their impairment is a major contributor to social and functional disability.

There is compelling evidence from recent meta-analyses that psychosocial approaches to cognitive remediation are effective in SZ. We have shown that a psychosocial cognitive rehabilitation known as Cognitive Enhancement Therapy (CET) substantially improves both social cognition and employment rates among patients with early course SZ. The effects were durable at 1 year following end of treatment.

CET is a comprehensive, developmental approach to address social and non-social cognitive deficits in SZ; it seeks to facilitate the development of adult social-cognitive milestones (e.g., perspective-taking, social context appraisal) by shifting thinking from reliance on effortful, serial processing to a "gistful" and spontaneous abstraction of social themes (details about CET in section C.2.6). CET targets social-cognitive impairments in perspective-taking and emotion regulation through computerized training in basic neurocognitive processes, and the use of social-cognitive rehabilitation groups. The efficacy of CET for remediating social-cognitive impairments in perspective-taking and emotion regulation in SZ presumably reflects an underlying change in fronto-temporal brain function and connectivity during the course of treatment, made possible by the plasticity of the human brain. CET may also protect against gray matter loss, and even support fronto-temporal gray matter growth in service of social-cognitive enhancement in SZ.

In this study, we plan to modify CET for individuals at CHR. We will develop a manual for CLUES and systematically test the acceptability, tolerability, adherence and preliminary proof of target engagement (part 1), and preliminary efficacy in a proof of concept open label trial (part 2). An important recent initiative in treatment development is to ensure informed, data-driven decisions early in clinical trials, i.e. to identify therapeutic targets, obtain evidence of target engagement and a proof of concept of efficacy prior to proceeding to expensive clinical trials. To pursue this goal, we will evaluate CET effects on cognition and social cognition in part 1 before efficacy testing in part 2.

Overview:

This study will be organized in two parts:

Part 1: Preliminary open-label CLUES group (n=8) to verify target engagement (using cognition and social cognition measures), to evaluate feasibility and tolerability, and to iteratively refine the manual.

Part 2: Small, randomized trial comparing CLUES (2 groups, n=15 each to a control condition (psychotherapy + an active computer-based program, Sporcle, with simple/ non-demanding computer games).CLUES Interventions in this part will be optimized based on part 1 results.

Interventions:

1) Individualized assessment: The intervention begins with a comprehensive assessment of neurocognition and social cognition, as well as cognitive style. This informs development of an individualized coaching plan targeting the individual's areas of difficulty. The individualized coaching plan sets CET apart from other more standardized cognitive remediation approaches. 2) Neurocognitive remediation sessions. Weekly CET cognitive remediation sessions involve working with a partner (peer) and is facilitated by a clinician. This provides a unique opportunity for participants to complete "bottom up" cognitive exercises designed to improve processing speed, attention, memory and problem solving while also learning to negotiate the social tasks involved in working with a partner (e.g., making appropriate small talk, paying attention and keeping score while a partner engages in the tasks, providing encouragement when a partner struggles, and/or managing feelings that come up when the participant struggles more than their partner). 3) Social cognitive group: Participants take part in weekly social cognitive groups concurrently with neurocognitive training and individual sessions. This group is designed to help participants learn strategies for applying skills to improve non-social and social cognition and provide in vivo learning experiences to foster the development of social wisdom and interpersonal success. A broad, theoretically-driven array of social-cognitive abilities are targeted in the social cognitive groups, which range from abstracting the "gist" or main point in social interactions to perspective taking, social context appraisal, and emotion management. Participants actively engage in the social cognitive groups by responding to unrehearsed social exchanges, presenting homework, participating in cognitive exercises that focus on experiential learning, providing feedback to peers, and chairing homework sessions. 4) Individual coaching: Weekly individual coaching sessions provide opportunities for the intervention to be further tailored to the participants' specific goals, cognitive difficulties and cognitive style. Coaching sessions help the participant to develop a training plan, digest information and skills learned in social cognitive group and in the neurocognitive training sessions, and figure out how to apply them to make progress toward personal goals.

Control treatment (Part 2 only):

During part 1, all participants will take part in CLUES. During part 2, we will conduct a small randomized trial in which participants will be randomized to CLUES or the control intervention (n=15 each). The control intervention will consist of weekly supportive personal therapy plus 2 hours/ week of participation in Sporcle, a web-based, publicly available active computer-based, generic, quiz-type program. Sporcle provides quizzes on subject areas from geography to basic arithmetic to pop-culture. Sporcle includes games such as identifying popular logos, naming as many pictured fruits and vegetables as possible, and listing state capitols. Based on online user data and on level of difficulty, relatively easy exercises are chosen (averaging approximately 70% accuracy (i.e. 70% of quiz items correctly answered, on average). Games are presented to participants on "prescription cards" each week, with an aim of participating in 2 hours per week (equivalent to 1 hour of lumosity plus 1 hour per week paired computer training.

In ST, patients meet individually with a therapist to learn and practice a variety of stress-reduction and illness management techniques. The ST approach is designed to be sensitive to the patient's stage of development and divided into 2 phases. The first, basic phase (0-3 months) focuses on psychoeducation about risk for psychosis (to be developed during phase 1), the role of stress in the disorder, and symptom exacerbation, and introduces basic coping strategies to minimize and/or avoid stress in one's life.The second, phase (4-6 months) advances to a personalized approach to the identification of early cues of distress and the application of healthy coping strategies to enhance adjustment. By tailoring the treatment to the patient's stage of recovery, Patients meet weekly with a therapist, although more frequent sessions are available if needed. We will seek to match the number of sessions or hours of treatment between CLUES and ST.

Participants will be assessed at: 1) Baseline, 2) 3 months into the program, 3) at the time of completion of the program (6 months), and 4) 3 months following completion of CLUES, in the part 2 trial only (Table 1). All these assessments will be administered during part 1 to assess acceptability, applicability to the CHR population and assessment burden; Observations will then be used to optimize assessment battery for part 2.

ELIGIBILITY:
Inclusion Criteria:

Broad criteria for clinical high risk for psychosis including meeting for SIPS clinical high risk syndrome or any two of the following:

* Trait risk: Having a first degree relative with a psychotic disorder, or a schizotypal disorder in the patient
* Positive symptoms: One or more of the attenuated SOPS Positive or Disorganized items scoring mild (3), moderate (4) or severe (5) but not at a psychotic level; these may include one or more Basic Symptoms (Klosterkotter et al 2001).
* Negative symptoms: Two or more of the SOPS negative symptoms rated at least moderate in severity
* Cognition: executive cognitive impairment (at least 1.0 standard deviation deficit relative to age-expected norms on at least 30% of the measures
* Functioning: GAF decline > 30% over the last 2 years, sustained for > 1 mo.

Exclusion Criteria:

* History of meeting full criteria for psychotic disorder
* Significant neurological or medical disorders that may produce cognitive impairment (e.g., seizure disorder, traumatic brain injury)
* More than 6 months (lifetime) of exposure to antipsychotic treatment
* A recent (within the past 3 months) history of substance abuse or dependence
* IQ < 80
* Failure to achieve at least a 6th grade reading level
* Persistent suicidal or homicidal behavior

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2015-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Social and Role Functioning at 6 Month and 9 Month (clinical interview) | Baseline, 6 month, and 9 month
  Assessed through clinical interview

SECONDARY OUTCOMES:
Change from Baseline in Neurocognitive functioning (neuropsychological test battery) | Baseline, 6 month, and 9 month
  Assessed through administration of neuropsychological test battery
Change from Baseline in Social-cognitive functioning (neuropsychological test battery) | Baseline, 6 month, and 9 month
  Assessed through administration of neuropsychological test battery
Satisfaction with treatment (Self report of client satisfaction) | 6 month and 9 months
  Self report of client satisfaction
Feasibility of treatment (Rates of attendance for all aspects of treatment) | 6 months and 9 months
  Rates of attendance for all aspects of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Matcheri Keshavan, MD, Principal Investigator — Beth Israel Deaconess Medical Center/ Massachusetts Mental Health Center
Locations (1):
- Beth Israel Deaconess Medical Center/ Massachusetts Mental Health Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Addington J, Cadenhead KS, Cannon TD, Cornblatt B, McGlashan TH, Perkins DO, Seidman LJ, Tsuang M, Walker EF, Woods SW, Heinssen R; North American Prodrome Longitudinal Study. North American Prodrome Longitudinal Study: a collaborative multisite approach to prodromal schizophrenia research. Schizophr Bull. 2007 May;33(3):665-72. doi: 10.1093/schbul/sbl075. Epub 2007 Jan 25. PMID 17255119
- [Background] Ben-Yishay Y, Piasetsky EB, Rattok J. A systematic method for ameliorating disorders in basic attention. In: Meir MJ, Benton AL, Diller L, eds. Neuropsychological Rehabilitation. New York, NY: Guilford; 1985:165 181.
- [Background] Bracy OL.PSSCogRehab.Indianapolis, IN: Psychological Software Services Inc; 1994.
- [Background] Cannon TD, Cadenhead K, Cornblatt B, Woods SW, Addington J, Walker E, Seidman LJ, Perkins D, Tsuang M, McGlashan T, Heinssen R. Prediction of psychosis in youth at high clinical risk: a multisite longitudinal study in North America. Arch Gen Psychiatry. 2008 Jan;65(1):28-37. doi: 10.1001/archgenpsychiatry.2007.3. PMID 18180426
- [Background] Cannon-Spoor HE, Potkin SG, Wyatt RJ. Measurement of premorbid adjustment in chronic schizophrenia. Schizophr Bull. 1982;8(3):470-84. doi: 10.1093/schbul/8.3.470. PMID 7134891
- [Background] Carrion RE, McLaughlin D, Goldberg TE, Auther AM, Olsen RH, Olvet DM, Correll CU, Cornblatt BA. Prediction of functional outcome in individuals at clinical high risk for psychosis. JAMA Psychiatry. 2013 Nov;70(11):1133-42. doi: 10.1001/jamapsychiatry.2013.1909. PMID 24006090
- [Background] Eack SM, Greenwald DP, Hogarty SS, Cooley SJ, DiBarry AL, Montrose DM, Keshavan MS. Cognitive enhancement therapy for early-course schizophrenia: effects of a two-year randomized controlled trial. Psychiatr Serv. 2009 Nov;60(11):1468-76. doi: 10.1176/appi.ps.60.11.1468. PMID 19880464
- [Background] Eack SM, Hogarty GE, Greenwald DP, Hogarty SS, Keshavan MS. Cognitive enhancement therapy improves emotional intelligence in early course schizophrenia: preliminary effects. Schizophr Res. 2007 Jan;89(1-3):308-11. doi: 10.1016/j.schres.2006.08.018. Epub 2006 Oct 19. PMID 17055227
- [Background] Eack SM, Hogarty GE, Cho RY, Prasad KM, Greenwald DP, Hogarty SS, Keshavan MS. Neuroprotective effects of cognitive enhancement therapy against gray matter loss in early schizophrenia: results from a 2-year randomized controlled trial. Arch Gen Psychiatry. 2010 Jul;67(7):674-82. doi: 10.1001/archgenpsychiatry.2010.63. Epub 2010 May 3. PMID 20439824
- [Background] Eack SM, Greeno CG, Pogue-Geile MF, Newhill CE, Hogarty GE, Keshavan MS. Assessing social-cognitive deficits in schizophrenia with the Mayer-Salovey-Caruso Emotional Intelligence Test. Schizophr Bull. 2010 Mar;36(2):370-80. doi: 10.1093/schbul/sbn091. Epub 2008 Jul 22. PMID 18648021
- [Background] Eack SM, Greenwald DP, Hogarty SS, Keshavan MS. One-year durability of the effects of cognitive enhancement therapy on functional outcome in early schizophrenia. Schizophr Res. 2010 Jul;120(1-3):210-6. doi: 10.1016/j.schres.2010.03.042. Epub 2010 May 15. PMID 20472402
- [Background] Eack SM, Hogarty GE, Greenwald DP, Hogarty SS, Keshavan MS. Effects of Cognitive Enhancement Therapy on Employment Outcomes in Early Schizophrenia: Results From a Two-Year Randomized Trial. Res Soc Work Pract. 2011 Jan 27;21(1):32-42. doi: 10.1177/1049731509355812. PMID 23885163
- [Background] Fisher M, Loewy R, Hardy K, Schlosser D, Vinogradov S. Cognitive interventions targeting brain plasticity in the prodromal and early phases of schizophrenia. Annu Rev Clin Psychol. 2013;9:435-63. doi: 10.1146/annurev-clinpsy-032511-143134. Epub 2013 Jan 7. PMID 23297786
- [Background] Fusar-Poli P, Borgwardt S, Bechdolf A, Addington J, Riecher-Rossler A, Schultze-Lutter F, Keshavan M, Wood S, Ruhrmann S, Seidman LJ, Valmaggia L, Cannon T, Velthorst E, De Haan L, Cornblatt B, Bonoldi I, Birchwood M, McGlashan T, Carpenter W, McGorry P, Klosterkotter J, McGuire P, Yung A. The psychosis high-risk state: a comprehensive state-of-the-art review. JAMA Psychiatry. 2013 Jan;70(1):107-20. doi: 10.1001/jamapsychiatry.2013.269. PMID 23165428
- [Background] Giuliano AJ, Li H, Mesholam-Gately RI, Sorenson SM, Woodberry KA, Seidman LJ. Neurocognition in the psychosis risk syndrome: a quantitative and qualitative review. Curr Pharm Des. 2012;18(4):399-415. doi: 10.2174/138161212799316019. PMID 22239571
- [Background] Green MF, Kern RS, Braff DL, Mintz J. Neurocognitive deficits and functional outcome in schizophrenia: are we measuring the "right stuff"? Schizophr Bull. 2000;26(1):119-36. doi: 10.1093/oxfordjournals.schbul.a033430. PMID 10755673
- [Background] Green MF, Hellemann G, Horan WP, Lee J, Wynn JK. From perception to functional outcome in schizophrenia: modeling the role of ability and motivation. Arch Gen Psychiatry. 2012 Dec;69(12):1216-24. doi: 10.1001/archgenpsychiatry.2012.652. PMID 23026889
- [Background] Heinrichs RW, Zakzanis KK. Neurocognitive deficit in schizophrenia: a quantitative review of the evidence. Neuropsychology. 1998 Jul;12(3):426-45. doi: 10.1037//0894-4105.12.3.426. PMID 9673998
- [Background] Hogarty GE, Flesher S, Ulrich R, Carter M, Greenwald D, Pogue-Geile M, Kechavan M, Cooley S, DiBarry AL, Garrett A, Parepally H, Zoretich R. Cognitive enhancement therapy for schizophrenia: effects of a 2-year randomized trial on cognition and behavior. Arch Gen Psychiatry. 2004 Sep;61(9):866-76. doi: 10.1001/archpsyc.61.9.866. PMID 15351765
- [Background] Hogarty, G. E., & Greenwald, D. P: Cognitive Enhancement Therapy: The Training Manual. University of Pittsburgh Medical Center: Authors. Available through www.CognitiveEnhancementTherapy.com, 2006.
- [Background] Keshavan MS, DeLisi LE, Seidman LJ. Early and broadly defined psychosis risk mental states. Schizophr Res. 2011 Mar;126(1-3):1-10. doi: 10.1016/j.schres.2010.10.006. Epub 2010 Nov 30. PMID 21123033
- [Background] Keshavan MS, Hogarty GE. Brain maturational processes and delayed onset in schizophrenia. Dev Psychopathol. 1999 Summer;11(3):525-43. doi: 10.1017/s0954579499002199. PMID 10532623
- [Background] Kohler CG, Turner TH, Bilker WB, Brensinger CM, Siegel SJ, Kanes SJ, Gur RE, Gur RC. Facial emotion recognition in schizophrenia: intensity effects and error pattern. Am J Psychiatry. 2003 Oct;160(10):1768-74. doi: 10.1176/appi.ajp.160.10.1768. PMID 14514489
- [Background] Mayer JD, Salovey P, Caruso DR, Sitarenios G. Measuring emotional intelligence with the MSCEIT V2.0. Emotion. 2003 Mar;3(1):97-105. doi: 10.1037/1528-3542.3.1.97. PMID 12899321
- [Background] McDonald S, Bornhofen C, Shum D, Long E, Saunders C, Neulinger K. Reliability and validity of The Awareness of Social Inference Test (TASIT): a clinical test of social perception. Disabil Rehabil. 2006 Dec 30;28(24):1529-42. doi: 10.1080/09638280600646185. PMID 17178616
- [Background] McGorry PD, Yung AR, Phillips LJ, Yuen HP, Francey S, Cosgrave EM, Germano D, Bravin J, McDonald T, Blair A, Adlard S, Jackson H. Randomized controlled trial of interventions designed to reduce the risk of progression to first-episode psychosis in a clinical sample with subthreshold symptoms. Arch Gen Psychiatry. 2002 Oct;59(10):921-8. doi: 10.1001/archpsyc.59.10.921. PMID 12365879
- [Background] Mesholam-Gately RI, Giuliano AJ, Goff KP, Faraone SV, Seidman LJ. Neurocognition in first-episode schizophrenia: a meta-analytic review. Neuropsychology. 2009 May;23(3):315-36. doi: 10.1037/a0014708. PMID 19413446
- [Background] Nuechterlein KH, Barch DM, Gold JM, Goldberg TE, Green MF, Heaton RK. Identification of separable cognitive factors in schizophrenia. Schizophr Res. 2004 Dec 15;72(1):29-39. doi: 10.1016/j.schres.2004.09.007. PMID 15531405
- [Background] Nuechterlein KH, Green MF, Kern RS, Baade LE, Barch DM, Cohen JD, Essock S, Fenton WS, Frese FJ 3rd, Gold JM, Goldberg T, Heaton RK, Keefe RS, Kraemer H, Mesholam-Gately R, Seidman LJ, Stover E, Weinberger DR, Young AS, Zalcman S, Marder SR. The MATRICS Consensus Cognitive Battery, part 1: test selection, reliability, and validity. Am J Psychiatry. 2008 Feb;165(2):203-13. doi: 10.1176/appi.ajp.2007.07010042. Epub 2008 Jan 2. PMID 18172019
- [Background] Waber DP, Holmes JM. Assessing children's copy productions of the Rey-Osterrieth Complex Figure. J Clin Exp Neuropsychol. 1985 Jun;7(3):264-80. doi: 10.1080/01688638508401259. PMID 3998091
- [Background] Wood SJ, Yung AR, McGorry PD, Pantelis C. Neuroimaging and treatment evidence for clinical staging in psychotic disorders: from the at-risk mental state to chronic schizophrenia. Biol Psychiatry. 2011 Oct 1;70(7):619-25. doi: 10.1016/j.biopsych.2011.05.034. Epub 2011 Jul 18. PMID 21762875
- [Background] Woodberry KA, Giuliano AJ, Seidman LJ. Premorbid IQ in schizophrenia: a meta-analytic review. Am J Psychiatry. 2008 May;165(5):579-87. doi: 10.1176/appi.ajp.2008.07081242. Epub 2008 Apr 15. PMID 18413704
- [Background] Vinogradov S, Fisher M, de Villers-Sidani E. Cognitive training for impaired neural systems in neuropsychiatric illness. Neuropsychopharmacology. 2012 Jan;37(1):43-76. doi: 10.1038/npp.2011.251. Epub 2011 Nov 2. PMID 22048465
- [Background] Wykes T, Huddy V, Cellard C, McGurk SR, Czobor P. A meta-analysis of cognitive remediation for schizophrenia: methodology and effect sizes. Am J Psychiatry. 2011 May;168(5):472-85. doi: 10.1176/appi.ajp.2010.10060855. Epub 2011 Mar 15. PMID 21406461